CLINICAL TRIAL: NCT06339723
Title: Examination of the Effectiveness of Training Given to Caregivers About Percutaneous Endoscopic Gastrostomy Using the Pecha Kuka Method to Caregivers Who Care for Palliative Care Patients
Brief Title: Pecha Kuka Method About Percutaneous Endoscopic Gastrostomy for Caregivers Who Care for Palliative Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024/03-17
Record Dates: First submitted 2024-02-23; First posted 2024-04-01 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Pecha Kuka; Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Training Given with the Pecha Kucha Method
  Interventions: Behavioral: Pecha Kucha
- Control (No Intervention): No training was given on the Pecha Kucha Method

INTERVENTIONS:
Behavioral: Pecha Kucha — Pecha Kucha Method training was given
  Arms: Experimental

SUMMARY:
Palliative care; It was started by Dame Cicely Saunders in the 1960s as a hospice for community-based provision. Today, palliative care is defined as care that begins with the patient's diagnosis, symptom management is carried out effectively, and a comprehensive, supportive, humanistic approach is based on the individual and his family. When the literature was examined, no study was found that evaluated the effectiveness of the training given by the Pecha Kuka method to caregivers caring for palliative care patients about percutaneous endoscopic gastrostomy. In addition, it is thought that the results of this research will shed light on identifying problems related to feeding practices in patients fed with PEG tubes and identifying misinformation and practices of caregivers. Determining the knowledge level and initiatives of caregivers regarding percutaneous endoscopic gastrostomy tube feeding practices will contribute to the development of educational activities and effective strategies. Study results may provide important data regarding improving the quality of care given to patients and caregivers after discharge and controlling complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Accepting research
* Being a relative of a palliative care patient
* Ability to communicate adequately

Exclusion Criteria:

* The patient's relative has a disability (such as vision, speech and hearing) that prevents them from communicating.
* No psychiatric problems

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Evaluation Form for Feeding Practices with Percutaneous Endoscopic Gastrostomy Tube: | 4 week
  This data collection tool was created by researchers to evaluate the nutritional practices of individuals caring for patients fed through PEG tubes. Storage of the enteral nutrition product, duration of use after opening, dressing the feeding tube, rotating the plate 360 degrees during dressing, positioning the patient during feeding, checking the number written at the entrance of the feeding tube every time the nutritional product is given to the patient, use of nutritional products, duration of administration of the enteral nutrition product
Visual Analog Scale -Anxiety: | 4 week
  Developed by Cline et al. It consists of a horizontal line 10 cm long. The left side contains the labels "no anxiety" and the right side includes the labels "I feel a lot of anxiety". The VAS value is determined by measuring the distance between the leftmost tip of the scale and the marked point. Values range from 0 to 10, with higher values indicating increased anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No